CLINICAL TRIAL: NCT02046655
Title: Corifollitropin Alfa Compared to Daily Rec FSH in Poor Responders Undergoing ICSI Using a GnRH Antagonist Protocol
Brief Title: Corifollitropin Alfa Compared to Daily rFSH in Poor Responders Undergoing ICSI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, E.M. Kolibianakis, Assistant Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHR-11
Record Dates: First submitted 2013-12-18; First posted 2014-01-28 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Subfertility
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Corifollitropin alfa group (Experimental): On day 2 of the cycle, a single subcutaneous (SC) dose of 150 μg Corifollitropin alfa (Elonva) will be administered.
  GnRH antagonist (Orgalutran) 0.25 mg/day flexible initiation by a follicle of 14mm.
  A daily dose of recFSH (450 IU/day) will be used from day 8 of stimulation until the day of hCG, if necessary.
  Triggering of final oocyte maturation will be performed using 250 μg of rechCG.
  Interventions: Drug: Corifollitropin alfa
- rec FSH group (Active Comparator): On day 2 of the cycle, daily SC dose of min 450 IU recFSH (Puregon) will be administered.
  GnRH antagonist (Orgalutran) 0.25 mg/day , flexible initiation by a follicle of 14mm.
  Triggering of final oocyte maturation will be performed using 250 μg of rechCG.
  Interventions: Drug: rFSH

INTERVENTIONS:
Drug: Corifollitropin alfa
  Other Names: Elonva
  Arms: Corifollitropin alfa group
Drug: rFSH
  Other Names: Puregon
  Arms: rec FSH group

SUMMARY:
Corifollitropin alfa has been shown to result in significantly more oocytes compared to daily recombinant follicle stimulating hormone (recFSH) (Devroey et al., 2009), probably due to the higher circulating FSH activity during the first days of stimulation. For this reason, the use of corifollitropin alfa might be beneficial in poor responders in whom the number of oocytes retrieved is crucial for success.

The purpose of this study is to evaluate the effectiveness of corifollitropin alfa treatment compared to daily recFSH in terms of the number of oocytes retrieved in a defined population of poor responder patients undergoing intracytoplasmic sperm injection (ICSI) using gonadotrophin releasing hormone (GnRH) antagonists.

ELIGIBILITY:
Inclusion Criteria:

1. Proven poor responders of couples with an indication for COS
2. ≥ 18 and < 45 years of age
3. BMI ≥ 18 and ≤ 32 kg/m2
4. Regular spontaneous menstrual cycle (24-35 days)
5. Availability of ejaculatory sperm (use of donated and/or cryo-preserved sperm is allowed)

Exclusion Criteria:

1. PGD or PGS
2. TESE

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Total number of retrieved oocytes | 36 h after human chorionic gonadotrophin (hCG) administration

SECONDARY OUTCOMES:
Clinical pregnancy rate (evidence of intrauterine sac with fetal heart activity at 6-8 weeks of gestation) | At 6-8 weeks of gestation
Number of embryos transferred | 2 days following oocyte retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Efstratios M Kolibianakis, MD, MSc, PhD, Principal Investigator — Unit for Human Reproduction, 1st Dept. of Obstetrics and Gynaecology, Medical School, Aristotle University of Thessaloniki
Locations (1):
- Unit for Human Reproduction, 1st Dept of Obstetrics and Gynaecology, Medical School, Aristotle University of Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Derived] Kolibianakis EM, Venetis CA, Bosdou JK, Zepiridis L, Chatzimeletiou K, Makedos A, Masouridou S, Triantafillidis S, Mitsoli A, Tarlatzis BC. Corifollitropin alfa compared with follitropin beta in poor responders undergoing ICSI: a randomized controlled trial. Hum Reprod. 2015 Feb;30(2):432-40. doi: 10.1093/humrep/deu301. Epub 2014 Dec 9. PMID 25492411